CLINICAL TRIAL: NCT07285928
Title: Contribution of Cerebral Pulsatility Assessment by Transcranial Ultrasound to the Decision-making for Cerebrospinal Fluid Shunting in Patients With Suspected Idiopathic Normal Pressure Hydrocephalus: a Prospective Cohort Study
Brief Title: Transcranial Ultrasound Assessment of Cerebral Pulsatility in Shunt Decision-making for Suspected Idiopathic Normal Pressure Hydrocephalus: a Prospective Cohort Study
Acronym: HYDROPULSE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR250159 - HYDROPULSE
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Brain Pulsatility; Idiopathic Normal Pressure Hydrocephalus (INPH)
Keywords: transcranial ultrasound; cerebral pulsatility; idiopathic normal pressure hydrocephalus (iNPH),

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients improved after CSF shunting surgery
- patients not improved after CSF shunting surgery

SUMMARY:
This will be a single-center, prospective, analytical cohort study. All included patients will undergo transcranial ultrasound (TPI) with measurement of cerebral pulsatility parameters prior to subtractive lumbar puncture during hospitalization in the neurosurgery department, followed by a second ultrasound assessment either at one year after surgery for operated patients, or at one year after the initial ultrasound assessment for non-operated patients. This ultrasound evaluation will be integrated into the routine work-up, which is already systematically performed in cases of suspected idiopathic normal pressure hydrocephalus (iNPH).

The neurosurgical team's decision to perform cerebrospinal fluid (CSF) shunting will be made blinded to the ultrasound measurements and based solely on the standard clinical protocol.

The primary objective of the study is to demonstrate that the mean amplitude of cerebral pulsatility (MeanBTP) prior to subtractive lumbar puncture is significantly higher in patients who show clinical improvement 12 months after CSF shunting compared with those who do not, with a type I error risk (alpha) of 0.05."

DETAILED DESCRIPTION:
This will be a prospective, single-center cohort study including patients with suspected idiopathic normal pressure hydrocephalus (iNPH). Eligibility will require fulfillment of inclusion criteria and confirmation of non-opposition after written informed consent procedures.

All patients will undergo transcranial pulse imaging (TPI) with measurement of cerebral pulsatility parameters prior to subtractive lumbar puncture during hospitalization. Operated patients will have a second TPI assessment at 12 months post-surgery, while non-operated patients will undergo repeat TPI 12 months after baseline. Ultrasound assessments will be integrated into the standard hydrocephalus work-up.

The decision to perform cerebrospinal fluid (CSF) shunting will be made by the neurosurgical team blinded to ultrasound findings and based solely on standard clinical and radiological criteria. Baseline clinical (demographics, vascular risk factors, cognitive/gait/urinary symptoms, neurological history) and radiological variables (ventricular volume, Evans index, callosal angle, DESH, Radscale) will be collected.

During hospitalization, gait and cognitive function will be evaluated before and 48 hours after lumbar puncture. TPI will provide two indices of cerebral pulsatility: mean brain tissue pulsatility (MeanBTP) and maximal brain tissue pulsatility (MaxBTP), expressed as peak amplitude, peak amplitude mean, and root mean square.

Follow-up will include standardized clinical and radiological assessments. Non-operated patients will be evaluated at 12 months. Operated patients will be seen at 2 months and 12 months postoperatively, with documentation of complications, shunt valve settings, ventricular volume changes, and subdural collections.

Statistical analyses will be performed using STATA v11 (StataCorp, USA). Continuous variables will be expressed as means ± SD or medians; categorical variables as percentages. Normality will be assessed with the Kolmogorov-Smirnov test, and variance equality with F-test. Comparisons will use Student's t-test, chi-square, or Fisher's exact test as appropriate. Cox proportional hazards regression will be applied for multivariable analysis. P < 0.05 will be considered significant.

The primary objective will be to demonstrate that the mean amplitude of cerebral pulsatility (MeanBTP) measured prior to subtractive lumbar puncture will be significantly higher in patients who show clinical improvement 12 months after cerebrospinal fluid (CSF) shunting compared with those who do not, with a type I error risk (alpha) of 0.05.

The secondary objectives will be to correlate cerebral pulsatility (measured by transcranial pulse imaging, TPI) with functional indices of iNPH and CSF shunting outcomes, including: speech therapy evaluation, physiotherapy-based gait assessment, global neurological disability, ventricular volume, and shunt valve opening pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Suspected iNPH (= at least 1/3 of the triad symptoms + ventriculomegaly on brain imaging)
* Hospitalised at Tours University Hospital for 'hydrocephalus assessment'
* Patient who has provided written and signed consent

Non-inclusion criteria

* Individuals who objected to data processing
* Walking assessment by the physiotherapy team impossible AND cognitive assessment by the speech therapy team impossible

Exclusion criteria

* Patients already fitted with a CSF shunting system (VPS)
* Suspicion of obstructive hydrocephalus (aqueduct stenosis, tumour, etc.)
* Patients under legal protection (guardianship, curatorship, judicial protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with suspected iNPH, hospitalized at Tours University Hospital for "hydrocephalus assessment"
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 12 months
  Clinical improvement at 12 months in patients who undergo CSF shunt surgery (ventriculoperitoneal shunt, VPS).
  Clinical improvement will be defined as cognitive improvement at 12 months and/or gait improvement at 12 months.
  * Cognitive improvement: improvement in at least two cognitive tests. Improvement in a single test will be defined as an increase ≥ 1 standard deviation between the baseline pre-lumbar puncture (pre-LP) speech therapy evaluation and the 12-month postoperative assessment.
  * Gait improvement: improvement in the Get Up and Go test and/or the 10-meter walk test (10MWT) between baseline and the 12-month postoperative assessment.

SECONDARY OUTCOMES:
Mattis Dementia Rating Scale score (MDRS) | 12 months
  Detailed speech therapy (neuropsychological) assessment: Mattis Dementia Rating Scale score (/144)
Wechsler Adult Intelligence Scale - 4th edition (WAIS-IV) | 12 months
  Detailed speech therapy (neuropsychological) assessment: WAIS-IV - Coding, Digit Span Forward, Digit Span Backward; Verbal fluency - literal and categorical; Trail Making Test A - duration (s) and errors; Rey-Osterrieth Complex Figure - copy duration (s) and copy score (/36); Rey Word List score (/15).
Get Up and Go test (s) | 12 months
  Detailed physiotherapy (motor) assessment: Get Up and Go test (s); Tinetti test (/28)
10-meter walk test | 12 months
  Detailed physiotherapy (motor) assessment: 10-meter walk test (10MWT) (s).
Reduction in modified Rankin Scale score (≤ 1 point compared with baseline) at 12 months | 12 months
  Global neurological disability assessment: modified Rankin Scale (/6).
Reduction in ventricular volume (total ventricular volume and third ventricular volume) at 12 months | 12 months
  Ventricular volume: measurement of total cerebral ventricular volume (mm³) and third ventricle volume (mm³) using a semi-automated technique with ITK-SNAP 4.2.0®.
Shunt valve opening pressure (mmH₂O) at 12 months | 12 months
  Shunt valve opening pressure: opening pressure value (mmH₂O) at 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ilyess ZEMMOURA, Pr, Principal Investigator — University Hospital, Tours
Locations (1):
- university hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ternifi R, Cazals X, Desmidt T, Andersson F, Camus V, Cottier JP, Patat F, Remenieras JP. Ultrasound measurements of brain tissue pulsatility correlate with the volume of MRI white-matter hyperintensity. J Cereb Blood Flow Metab. 2014 Jun;34(6):942-4. doi: 10.1038/jcbfm.2014.58. Epub 2014 Apr 9. PMID 24714033
- [Background] Byram B, Trahey GE, Palmeri M. Bayesian speckle tracking. Part II: biased ultrasound displacement estimation. IEEE Trans Ultrason Ferroelectr Freq Control. 2013 Jan;60(1):144-57. doi: 10.1109/TUFFC.2013.2546. PMID 23287921
- [Background] LANGFITT TW, KASSELL NF, WEINSTEIN JD. CEREBRAL BLOOD FLOW WITH INTRACRANIAL HYPERTENSION. Neurology. 1965 Aug;15:761-73. doi: 10.1212/wnl.15.8.761. No abstract available. PMID 14315301
- [Background] Kucewicz JC, Dunmire B, Giardino ND, Leotta DF, Paun M, Dager SR, Beach KW. Tissue pulsatility imaging of cerebral vasoreactivity during hyperventilation. Ultrasound Med Biol. 2008 Aug;34(8):1200-8. doi: 10.1016/j.ultrasmedbio.2008.01.001. Epub 2008 Mar 12. PMID 18336991
- [Background] Kucewicz JC, Dunmire B, Leotta DF, Panagiotides H, Paun M, Beach KW. Functional tissue pulsatility imaging of the brain during visual stimulation. Ultrasound Med Biol. 2007 May;33(5):681-90. doi: 10.1016/j.ultrasmedbio.2006.11.008. PMID 17346872
- [Background] Biogeau J, Desmidt T, Dujardin PA, Ternifi R, Eudo C, Vierron E, Remenieras JP, Patat F, Camus V, Constans T. Ultrasound Tissue Pulsatility Imaging Suggests Impairment in Global Brain Pulsatility and Small Vessels in Elderly Patients with Orthostatic Hypotension. J Stroke Cerebrovasc Dis. 2017 Feb;26(2):246-251. doi: 10.1016/j.jstrokecerebrovasdis.2016.09.002. Epub 2016 Nov 25. PMID 27894887
- [Background] Desmidt T, Hachemi ME, Remenieras JP, Lecomte P, Ferreira-Maldent N, Patat F, Camus V. Ultrasound Brain Tissue Pulsatility is decreased in middle aged and elderly type 2 diabetic patients with depression. Psychiatry Res. 2011 Jul 30;193(1):63-4. doi: 10.1016/j.pscychresns.2011.01.002. Epub 2011 May 17. PMID 21592742
- [Background] Eide PK, Brean A. Intracranial pulse pressure amplitude levels determined during preoperative assessment of subjects with possible idiopathic normal pressure hydrocephalus. Acta Neurochir (Wien). 2006 Nov;148(11):1151-6; discussion 1156. doi: 10.1007/s00701-006-0896-0. Epub 2006 Oct 16. PMID 17039303
- [Background] Eide PK. Intracranial pressure parameters in idiopathic normal pressure hydrocephalus patients treated with ventriculo-peritoneal shunts. Acta Neurochir (Wien). 2006 Jan;148(1):21-9; discussion 29. doi: 10.1007/s00701-005-0654-8. Epub 2005 Nov 14. PMID 16284706
- [Background] Eide PK, Sorteberg W. Diagnostic intracranial pressure monitoring and surgical management in idiopathic normal pressure hydrocephalus: a 6-year review of 214 patients. Neurosurgery. 2010 Jan;66(1):80-91. doi: 10.1227/01.NEU.0000363408.69856.B8. PMID 20023540
- [Background] Baroncini M, Baledent O, Ardi CE, Delannoy VD, Kuchcinski G, Duhamel A, Ares GS, Lejeune JP, Hodel J. Ventriculomegaly in the Elderly: Who Needs a Shunt? A MRI Study on 90 Patients. Acta Neurochir Suppl. 2018;126:221-228. doi: 10.1007/978-3-319-65798-1_45. PMID 29492565
- [Background] Bradley WG Jr, Scalzo D, Queralt J, Nitz WN, Atkinson DJ, Wong P. Normal-pressure hydrocephalus: evaluation with cerebrospinal fluid flow measurements at MR imaging. Radiology. 1996 Feb;198(2):523-9. doi: 10.1148/radiology.198.2.8596861.
- [Background] Stecco A, Cassara A, Zuccala A, Anoaica MB, Genovese E, Car PG, Panzarasa GP, Guzzardi G, Carriero A. Quantitative analysis of cerebrospinal fluid dynamics at phase contrast cine-MRI: predictivity of neurosurgical "Shunt" responsiveness in patients with idiopathic normal pressure hydrocephalus. J Neurosurg Sci. 2020 Oct;64(5):420-426. doi: 10.23736/S0390-5616.17.04092-9. Epub 2017 Sep 4. PMID 28869371
- [Background] Garcia-Armengol R, Domenech S, Botella-Campos C, Goncalves FJ, Menendez B, Teixidor P, Munoz-Narbona L, Rimbau J. Comparison of elevated intracranial pressure pulse amplitude and disproportionately enlarged subarachnoid space (DESH) for prediction of surgical results in suspected idiopathic normal pressure hydrocephalus. Acta Neurochir (Wien). 2016 Nov;158(11):2207-2213. doi: 10.1007/s00701-016-2858-5. Epub 2016 Jun 27. PMID 27349896
- [Background] Hamilton RB, Scalzo F, Baldwin K, Dorn A, Vespa P, Hu X, Bergsneider M. Opposing CSF hydrodynamic trends found in the cerebral aqueduct and prepontine cistern following shunt treatment in patients with normal pressure hydrocephalus. Fluids Barriers CNS. 2019 Jan 22;16(1):2. doi: 10.1186/s12987-019-0122-0. PMID 30665428
- [Background] Forner Giner J, Sanz-Requena R, Florez N, Alberich-Bayarri A, Garcia-Marti G, Ponz A, Marti-Bonmati L. Quantitative phase-contrast MRI study of cerebrospinal fluid flow: a method for identifying patients with normal-pressure hydrocephalus. Neurologia. 2014 Mar;29(2):68-75. doi: 10.1016/j.nrl.2013.02.016. Epub 2013 May 3. English, Spanish. PMID 23643684
- [Background] Craven CL, Toma AK, Mostafa T, Patel N, Watkins LD. The predictive value of DESH for shunt responsiveness in idiopathic normal pressure hydrocephalus. J Clin Neurosci. 2016 Dec;34:294-298. doi: 10.1016/j.jocn.2016.09.004. Epub 2016 Sep 28. PMID 27692614
- [Background] Kockum K, Virhammar J, Riklund K, Soderstrom L, Larsson EM, Laurell K. Diagnostic accuracy of the iNPH Radscale in idiopathic normal pressure hydrocephalus. PLoS One. 2020 Apr 24;15(4):e0232275. doi: 10.1371/journal.pone.0232275. eCollection 2020. PMID 32330190
- [Background] Yamada S, Ishikawa M, Yamamoto K. Optimal Diagnostic Indices for Idiopathic Normal Pressure Hydrocephalus Based on the 3D Quantitative Volumetric Analysis for the Cerebral Ventricle and Subarachnoid Space. AJNR Am J Neuroradiol. 2015 Dec;36(12):2262-9. doi: 10.3174/ajnr.A4440. Epub 2015 Sep 10. PMID 26359148
- [Background] Ishii K, Kanda T, Harada A, Miyamoto N, Kawaguchi T, Shimada K, Ohkawa S, Uemura T, Yoshikawa T, Mori E. Clinical impact of the callosal angle in the diagnosis of idiopathic normal pressure hydrocephalus. Eur Radiol. 2008 Nov;18(11):2678-83. doi: 10.1007/s00330-008-1044-4. Epub 2008 May 24. PMID 18500524
- [Background] Yamashita F, Sasaki M, Takahashi S, Matsuda H, Kudo K, Narumi S, Terayama Y, Asada T. Detection of changes in cerebrospinal fluid space in idiopathic normal pressure hydrocephalus using voxel-based morphometry. Neuroradiology. 2010 May;52(5):381-6. doi: 10.1007/s00234-009-0610-z. Epub 2009 Oct 22. PMID 19847409
- [Background] Ishii K, Kawaguchi T, Shimada K, Ohkawa S, Miyamoto N, Kanda T, Uemura T, Yoshikawa T, Mori E. Voxel-based analysis of gray matter and CSF space in idiopathic normal pressure hydrocephalus. Dement Geriatr Cogn Disord. 2008;25(4):329-35. doi: 10.1159/000119521. Epub 2008 Mar 5. PMID 18319598
- [Background] Sasaki M, Honda S, Yuasa T, Iwamura A, Shibata E, Ohba H. Narrow CSF space at high convexity and high midline areas in idiopathic normal pressure hydrocephalus detected by axial and coronal MRI. Neuroradiology. 2008 Feb;50(2):117-22. doi: 10.1007/s00234-007-0318-x. Epub 2007 Nov 9. PMID 17992524
- [Background] Miyajima M, Kazui H, Mori E, Ishikawa M; , on behalf of the SINPHONI-2 Investigators. One-year outcome in patients with idiopathic normal-pressure hydrocephalus: comparison of lumboperitoneal shunt to ventriculoperitoneal shunt. J Neurosurg. 2016 Dec;125(6):1483-1492. doi: 10.3171/2015.10.JNS151894. Epub 2016 Feb 12. PMID 26871203
- [Background] Carlsen JF, Munch TN, Hansen AE, Hasselbalch SG, Rykkje AM. Can preoperative brain imaging features predict shunt response in idiopathic normal pressure hydrocephalus? A PRISMA review. Neuroradiology. 2022 Nov;64(11):2119-2133. doi: 10.1007/s00234-022-03021-9. Epub 2022 Jul 24. PMID 35871239
- [Background] Nakajima M, Yamada S, Miyajima M, Ishii K, Kuriyama N, Kazui H, Kanemoto H, Suehiro T, Yoshiyama K, Kameda M, Kajimoto Y, Mase M, Murai H, Kita D, Kimura T, Samejima N, Tokuda T, Kaijima M, Akiba C, Kawamura K, Atsuchi M, Hirata Y, Matsumae M, Sasaki M, Yamashita F, Aoki S, Irie R, Miyake H, Kato T, Mori E, Ishikawa M, Date I, Arai H; research committee of idiopathic normal pressure hydrocephalus. Guidelines for Management of Idiopathic Normal Pressure Hydrocephalus (Third Edition): Endorsed by the Japanese Society of Normal Pressure Hydrocephalus. Neurol Med Chir (Tokyo). 2021 Feb 15;61(2):63-97. doi: 10.2176/nmc.st.2020-0292. Epub 2021 Jan 15. PMID 33455998
- [Background] Mori E, Ishikawa M, Kato T, Kazui H, Miyake H, Miyajima M, Nakajima M, Hashimoto M, Kuriyama N, Tokuda T, Ishii K, Kaijima M, Hirata Y, Saito M, Arai H; Japanese Society of Normal Pressure Hydrocephalus. Guidelines for management of idiopathic normal pressure hydrocephalus: second edition. Neurol Med Chir (Tokyo). 2012;52(11):775-809. doi: 10.2176/nmc.52.775. PMID 23183074
- [Background] Ishikawa M, Hashimoto M, Kuwana N, Mori E, Miyake H, Wachi A, Takeuchi T, Kazui H, Koyama H. Guidelines for management of idiopathic normal pressure hydrocephalus. Neurol Med Chir (Tokyo). 2008;48 Suppl:S1-23. doi: 10.2176/nmc.48.s1. PMID 18408356